CLINICAL TRIAL: NCT03783364
Title: Feasibility Study on Pre or Postoperative Accelerated Radiotherapy (POP-ART) in Breast Cancer Patients
Brief Title: Pre- or Postoperative Accelerated Radiotherapy
Acronym: POP-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC /2018/0996
Record Dates: First submitted 2018-10-05; First posted 2018-12-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Radiation Toxicity
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative (Experimental): preoperative radiotherapy
  Interventions: Radiation: Radiotherapy
- postoperative (Active Comparator): postoperative radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Pre- or postoperative acellerated irradition in 5 fractions

SUMMARY:
20 non-metastasized breast cancer patients receiving neoadjuvant chemotherapy will be randomized between preop or postop RT. Patients with clinically suspicious axillary lymph nodes will receive a fine needle biopsy. Patients receiving postop RT will receive neoadjuvant CT followed by surgery (21-28 days after CT) and adjuvant RT starting 28-35 days after surgery. Patients receiving preop RT will receive RT first, followed by CT (5-8 days after the end of RT) and surgery (21-28 days after CT). All patients will receive a clip to locate the tumor before the start of any treatment.

DETAILED DESCRIPTION:
In early-stage breast cancer the cornerstone of treatment is surgery. There are 2 possibilities: either mastectomy (ME, the whole breast, including the tumour, is removed) or breast-conserving surgery (BCS, only the tumour is removed, along with a part of the surrounding healthy tissue). After surgery, most patients also receive some kind of adjuvant systemic therapy like hormone therapy, chemotherapy (CT), targeted therapy or a combination of these. After BCS, adjuvant radiotherapy (RT) has shown to improve locoregional control and overall survival rates. After ME, a benefit of adjuvant RT was observed only in node positive patients. In recent years, adjuvant or postoperative (postop) CT is more and more replaced by preoperative (preop) or neo-adjuvant CT in patients with large tumours since the need for mastectomy may then be significantly decreased. Several randomized controlled trials demonstrated that there is no difference in overall survival whether CT is given pre- or postoperatively.

The use of breast RT in the neo-adjuvant setting is far less common. It has been proposed for patients with inoperable or inflammatory breast cancer and a recent retrospective study in breast cancer patients showed preop RT might improve disease free survival compared to postop RT. In another retrospective study comparing neoadjuvant versus adjuvant radio- and chemotherapy a possible benefit of neoadjuvant treatment was suggested for tumours larger than 2 cm. These benefits have also been observed in other cancer sites. There is evidence from randomized trials that preop RT is more effective than postop RT in patients with rectal carcinoma. For soft tissue sarcoma, better local control rates have been described with preop than with postop RT. From a radiobiological point of view, the benefits of giving RT preoperatively are not surprising. In contrast to the postop setting, the vasculature is still intact and less radioresistant tumour clones are present, both possibly increasing radiosensitivity. But there are other advantages of preop RT treatment. On the postop imaging used for RT planning, the localisation of the initial tumor is challenging, even with the aid of surgical clips. This is especially the case in patients receiving chemotherapy which is typically given before RT, thus increasing the interval between surgery and radiotherapy to about 6 months. In this 6-month period, tissue distortion and seroma, which are useful to guide the radiation oncologist when delineating the target volume for boost irradiation, have often disappeared. In the postop setting, larger volumes are delineated and interobserver variability is larger than in the preop setting. Preop breast irradiation has the advantage that the tumour is still in place and easy to locate. Zones of higher doses can be better targeted. For the latter reason, less acute side effects and a better overall breast cosmesis is expected. There is also a possibility of downsizing the tumour which might lead to a lower need for mastectomy. While preop breast RT clearly has some advantages, there are some obstacles that complicate its introduction into daily practice. One of these is the fear of delaying surgery and/or chemotherapy for too long. At Ghent University, investigators have experience with a 5-fraction RT schedule allowing preop RT delivery in a very short time span. Large randomized trials confirm that moderate hypofractionation schemes in 15 or 16 fractions are at least equivalent in tumor control and toxicity although the total dose is lower than the traditional 50 Gy in 25 fractions. Further acceleration to 5 fractions is expected to have an even greater radiobiological advantage concerning tumor control. In the UK FAST randomized trial, a schedule of 5 times 5.7 Gy, once a week, was compared to a normofractionation schedule of 25 times 2 Gy. Tumor control and toxicity were comparable after 3 years of follow-up. At Ghent University Hospital (UZ Gent) a feasibility trial was started using the FAST scheme (5 x 5.7 Gy) over 12 days (instead of 5 weeks) in patients of 65 years or older. Additionally, patients requiring a boost received a simultaneously integrated boost to the tumor bed of 5 x 6.5 Gy. The final analysis on 95 patients shows <10% grade 2-3 erythema, with only one case of moist desquamation, located at a skin fold(10). With this RT schedule of 5 fractions in 12 days given preoperatively, the investigators hypothesize that overall treatment time will not be increased.

The 3 main objectives of this project are: 1 - to prove the feasibility of preop breast RT in 5 fractions in patients also receiving neoadjuvant CT; 2 - to identify the involved cell death mechanisms and the effect of preop breast RT on the in-situ immune micro-environment; and 3 - to identify the markers that predict for response and toxicity.

Classically, radiotherapy is considered to mediate its effects via the direct killing of cancer cells. It is now known that radiotherapy can induce systemic effects resulting in tumour responses outside the irradiated regions. This phenomenon called the "abscopal"-effect has been reported in breast and several kinds of malignancies and is nowadays considered to be immune mediated. The hypothesis is that radiotherapy induces immunogenic cell death (ICD) through the release of tumour-associated antigens and damage associated molecular patterns (DAMPs), which leads to antigen uptake and dendritic cell maturation, resulting in the priming and clonal expansion of cytotoxic T-lymphocytes (CTLs) in the lymph nodes. These CTLs then travel back to the tumour, becoming tumour-infiltrating lymphocytes (TILs). Radiation could increase these TILs in a clinical setting and, more importantly, a high level of (post-therapy) TILs is associated with a good prognosis. Immunogenic cell death implicates the release of DAMPs and tumoral antigens through a disintegrated cell plasma membrane. The latter correlates with necrosis (regulated or secondary) instead of apoptosis, which was considered to be the principal mechanism of radiation induced cell death for years. Distinct cell death modalities may thus have a different (immunogenic) outcome. In this project the investigators would like to determine the mode of cell death evoked by high-dose pre-operative RT through measurement by immunohistochemistry (IHC) of cell death markers on pre-treatment, post-RT (only in case of pre-operative RT) as well as tumorectomy tissue samples. The investigators will correlate the results of the IHC stainings for cell death markers with the presence (or increase) of tumour infiltrating lymphocytes (TILs) in the same tissue samples and response to treatment. The number of TILs before and after radiotherapy will be assessed according to international guidelines.

Extracellular vesicles (EVs), such as exosomes (50-150 nm) are composed of a lipid bilayer that contains transmembrane proteins (such as receptors and adhesion molecules) derived from the donor cell and encloses soluble hydrophilic components derived from the cytosol of the donor cell such as signaling molecules, and nucleic acids (small RNAs such as miRNA). Different cell types can release EVs, including immune cells (monocytes, neutrophils, etc.), tumour cells, fibroblasts and adipocytes (fat cells). EVs are promising novel biomarkers because: 1) their molecular content is a fingerprint of the releasing cells and their status and consists of proteins, lipids, and nucleic acids, 2) they are released in easily accessible body fluids including blood and 3) they are enriched for highly selected biomarkers which otherwise would constitute only a very small proportion (less than 0.01%) of the total molecular content of blood. Analysis of Glypican-1 positive EVs in circulation distinguishes with absolute specificity and sensitivity healthy subjects and patients with a benign pancreatic disease from patients with early- and late-stage pancreatic cancer. EV transfer from stromal to breast cancer cells regulates therapy resistance pathways. miRNA levels in circulating EVs identify remnant vital tumour tissue and are suitable to measure therapy response and relapse monitoring. These pioneering studies suggest that quantification and characterization of EVs can be implemented to predict therapy response.

20 non-metastasized female breast cancer patients receiving neoadjuvant chemotherapy (CT) will be randomized between preop or postop RT. For each patient, a biopsy with tumor histology, histological grade, ER/PR status, Her2/Neu status (amplification or not) and Ki67 status will be available. Menopausal status will be assessed before the start of treatment. Patients with regular menses will be considered premenopausal. Patients > 50 years old with > 1 year of amenorrhea will be considered postmenopausal. In all other patients or patients with an intrauterine device or hysterectomy, plasma levels of LH, FSH and estradiol will be measured and documented.

Patients with clinically suspicious axillary lymph nodes will receive a fine needle biopsy. If lymph node involvement is confirmed by fine needle biopsy, they will receive an axillary clearance after neoadjuvant treatment and axillary RT will be performed (either preop or postop). In clinically node negative patients with a tumour of ≤ 5 cm, a sentinel node biopsy will be performed before the start of RT or CT. Patients with a tumour of > 5 cm, clinically node negative, will receive axillary clearance and axillary RT since a sentinel node biopsy is unreliable in these large tumours. Patients receiving postop RT will receive neoadjuvant CT followed by surgery (21-28 days after CT) and adjuvant RT starting 28-35 days after surgery. Patients receiving preop RT will receive RT first, followed by CT (5-8 days after the end of RT) and surgery (21-28 days after CT). All patients will receive a clip to locate the tumor before the start of any treatment.

The feasibility of preop RT will be evaluated based on overall treatment time. From a clinical point of view, it is not warranted that preop RT leads to an increase in the overall treatment time, since this may compromise locoregional control and survival. However, it is expected that preop RT will shorten the overall treatment time with about 14 days (SD 9 days) since the interval between RT and CT is shortened considerably. A difference of less than 14 days is not considered clinically relevant. With 20 patients (10 patients in every treatment arm), a 14 days' difference in overall treatment time can be detected with a power of > 90% (2-sided t-test, α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

All of the following inclusion criteria must be met:

* female patients with non-metastatic breast cancer,
* biopsy proven,
* age ≥ 18 years,
* WHO performance status 0 or 1,
* using contraceptives if in reproductive age category
* eligible for neo-adjuvant CT after multidisciplinary decision,
* informed consent obtained, signed and dated before specific protocol procedures.

Exclusion Criteria:

Any one or combination of the following:

* distant metastases,
* inflammatory breast cancer (mastitis carcinomatosa),
* multifocal tumor,
* lobular carcinoma,
* bilateral breast cancer,
* history of cancer, with the exception of non-melanoma skin cancer, in situ cervix carcinoma
* history of chemotherapy,
* history of radiation treatment,
* pregnant or breast feeding, or not using contraceptives if in reproductive age category
* exclusion criteria for chemotherapy:

  * leukocytes < 2500
  * absolute neutrophil count < 1000/µL
  * hemoglobine < 8 g/dL (transfusion is allowed)
  * platelets < 100 000/µl
  * total bilirubine > 1.5 x maximal normal reference range
  * AST > 2.5 x maximal normal reference range
  * ALT > 2.5 x maximal normal reference range
  * creatinine > 1.5 x maximal normal reference range
* Left ventricular ejection fraction (LVEF) < 55%
* planned immediate reconstructive surgery,
* conditions making toxicity evaluation difficult (e.g. skin disorders),
* Amiodarone treatment in the last 6 months
* patients unlikely to comply with the protocol (e.g. inability to return for follow-up visits or unlikely to complete the study).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of preop RT will be assessed in terms of overall treatment time | 4 years
  Treatment time will be measured.

SECONDARY OUTCOMES:
Breast symptoms: pain | 2 years
  none, only on contact, not only on contact, but occasionally, not only on contact and regularly, need for pain medication
Breast symptoms:Sense of heaviness | 2 years
  yes, no
Breast symptoms:Itching | 2 years
  none, occasionally, regularly
Arm symptoms: pain | 2 years
  none, occasionally, regularly
Arm symptoms: sense of heaviness | 2 years
  yes or no
Shoulder symptoms: pain | 2 years
  none, occasionally, regularly
Shoulder symptoms: Impaired mobility | 2 years
  yes, no
Pain other than breast, shoulder or arm pain | 2 years
  none, occasionally, regularly
Dysphagia according to the CTCAEE v. 4.03 | 2 years
  None; Symptomatic, able to eat regular diet; Symptomatic and altered eating/swallowing; Severely altered eating/swallowing; tube feeding or TPN or hospitalization indicated; Life-threatening consequences, urgent intervention indicated
Dyspnea according to the CTCAE v. 4.03 | 2 years
  None; Shortness of breath with moderate exertion; Shortness of breath with minimal exertion; limiting instrumental ADL; Shortness of breath at rest; limiting self-care ADL; Life-threatening consequences, urgent intervention indicated
Cough according to the CTCAE v. 4.03 | 2 years
  None, Mild symptoms, nonprescription intervention indicated, Moderate symptoms, medical intervention indicated; limiting instrumental ADL, Severe symptoms; limiting self-care ADL
Fatigue according to the CTCAE v. 4.03 | 2 years
  None; Fatigue relieved by rest; Fatigue not relieved by rest, limiting instrumental ADL; Fatigue not relieved by rest, limiting self-care ADL
Breast edema | 2 years
  none swelling or obscuration of anatomic architecture on close inspection Readily apparent obscuration of anatomic architecture, obliteration of skin folds; readily apparent deviation from normal anatomic contour, limiting instrumental ADL Gross deviation from normal anatomic contour, limiting self-care ADL
Dermatitis/desquamation according to the CTCAE v. 4.03 | 2 years
  none Faint erythema or dry desquamation Moderate to brisk erythema; moderate edema; patchy moist desquamation, mostly confined to skin folds and creases Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion2 Life-threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated
Desquamation | 2 years
  none dry desquamation moist desquamation
Troponine T value | 2 years
  in pg/ml
identify the involved cell death mechanisms and the effect of preop breast RT on the in-situ immune micro-environment | 3 years
  Liquid biopsies will be taken at fixed time points to search for biomarkers of response and toxicity. Chromatographic approaches combined with density gradient centrifugation is required to enrich EVs from plasma with minimal remnants of Argonaute-2 protein-miRNA complexes and high-density lipoproteins. Standard operating procedures have been optimized to enrich plasma EVs, to extract proteins/RNA and to perform proteomics/small RNA sequencing. EVs will be isolated following SOPs, quantified by nanoparticle tracking analysis and analysed by label free mass spectrometry and RNA sequencing. Receiver Operating Characteristics illustrate the performance of a biomarker, the sensitivity versus specificity, and will allow the selection of possible optimal EV biomarkers.
search for biomarkers of response and toxicity | 4 years
  To determine the mode of cell death evoked by pre-operative RT and its effect on the in-situ immune micro-environment measurement (by immunohistochemistry (IHC)) of cell death markers and TILs will be performed on pre-treatment, post-RT (only in case of pre-operative RT) as well as tumorectomy tissue samples. The results of the IHC stainings for cell death markers will be correlated with the presence (or increase) of TILs in the same tissue samples and response to treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Department of Radiotherapy, University Hospital Ghent, Ghent, Oost-Vlaanderen
  - University Hospital Ghent, Ghent